CLINICAL TRIAL: NCT05553067
Title: Oncogenic Role of Engrailed (EN)-2 in Epithelial Ovarian Neoplasms.
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Maisa Hashem Mohammed, Lecturer of Pathology, Sohag University
Other Study IDs: Soh-Med-22-09-13
Record Dates: First submitted 2022-09-21; First posted 2022-09-23 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Ovarian Neoplasms
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: Immunohistochemical staining of normal and neoplastic ovarian tissues by anti human Engrailed-2 antibody. — Immunohistochemical staining of normal and neoplastic ovarian tissues by anti human Engrailed-2 antibody and compare levels of expression in different ovarian specimens to detect its potential role in oncogenesis of ovarian carcinoma.

SUMMARY:
Detection of the potential oncogenic role of Engrailed-2 in epithelial ovarian neoplasms, in order to detect biological markers that could be targeted and blocked by new medications.

DETAILED DESCRIPTION:
Epithelial ovarian carcinomas represent more than 90% of all ovarian carcinomas. Treatment of these ovarian carcinomas on basis of their histopathological features didn't improve patients' outcomes with very high incidence of relapses and resistance to therapy. Detection of novel biological markers which are involved in tumor progression could have promising results if these biological molecules are targeted and blocked by new medications.

Engrailed-2 is a protein encoded by a gene located on chromosome 7. Engrailed-2 is involved in neural development and neural connections during embryological life. it has been proved that Engrailed-2 is expressed in non neural neoplasms, especially in prostatic and urinary bladder carcinomas. Now estimatiion of urinary and serum levels of Engrailed-2 is used as a non-invasive screening tool in to detect prostatic and urinary bladder carcinomas. We aim to evaluated immunohistochemical expression of Engrailed-2 in normal and neoplastic ovarian tissues and to compare such expression between normal and neoplastic tissues in order to improve its oncogenic role in ovarian carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* All types of epithelial ovarian neoplasms (benign, borderline and malignant).

Exclusion Criteria:

* Non-epithelial and/ or secondary ovarian tumors.
* Cases with poor clinical data.
* Cases who had history of pre-operative chemotherapy.

Ages: 20 Years to 70 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: This study will be applied on archived formalin-fixed, paraffin embedded ovarian tissue blocks from women who had ovarian benign, borderline and invasive malignant neoplasms and admitted to Obstetrics and Gynecology Department, Sohag University Hospital where they underwent oophorectomy operations because of benign and/ or malignant indications, from 2015 to 2021.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
compare levels of Engrailed-2 expression in different ovarian specimens. | December, 2021
  compare levels of immunohistochemical expression of Engrailed-2 in normal and neoplastic ovarian tissues. and correlate Engrailed-2 expression in neoplastic ovarian tissues to patients' ages, tumor phenotype and state of nodal metastasis.

CONTACTS AND LOCATIONS:
Overall Officials: Maisa H Mohammed, MD, Principal Investigator — Sohag University
Locations (1):
- Sohag faculty of medicine, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes
the participants will share the statistical analysis record and the informed consent form.
Supporting Information: SAP, ICF
Time Frame: within six months after publication.
Access Criteria: the principle investigator will share the statistical analysis record and the informed consent form on her account on research gate.
URL: https://www.researchgate.net/